CLINICAL TRIAL: NCT00593099
Title: A Preliminary Study of Sustained-Release Bupropion for Smoking Cessation in Bipolar Affective Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Tony P. George, M.D., FRPCP, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26254
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2007-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Nicotine Dependence; Smoking Cessation; Bupropion, sustained-release
MeSH Terms: conditions — Bipolar Disorder; Tobacco Use Disorder; Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Buproprion
  Interventions: Drug: Bupropion
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupropion — BUP [as the intermediate-release (IR) formulation] was inducted on Day 1 of the trial at 75 mg po qd x 3 days, then increased to 150 mg [as BUP SR formulation] qd x 4 days, and then increased to a final dose of up to 150 mg po bid (300 mg/day) by Day 15 (target quit date; TQD) as tolerated. This dose was continued for an additional eight (8) weeks at up to 150 mg po bid. Flexible dosing was permitted to allow for adjustments needed if a bipolar subject did not tolerate the full dose of BUP at 300 mg/day. BUP was discontinued at the end of Week 10.
  Other Names: Zyban
  Arms: 1
Drug: Placebo — matching placebo capsules (PLA) containing only a dextrose matrix.
  Arms: 2

SUMMARY:
The purpose of this pilot study is to determine the safety and potential efficacy of sustained-release bupropion (Zyban®) for the treatment of nicotine dependence in patients with bipolar affective illness. It is hypothesized that bupropion will produce a significant enhancement of smoking abstinence compared to placebo and will be safe for use in these patients.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the safety and potential efficacy of sustained-release bupropion (Zyban®) for the treatment of nicotine dependence in patients with bipolar affective illness. we propose to conduct a preliminary study of the safety and efficacy of bupropion SR (with flexible dosing up to 300 mg/day) in comparison to placebo in medication-maintained and stabilized outpatients with bipolar I and II disorder who are currently depressed despite mood-stabilizing medication and who are also nicotine-dependent cigarette smokers, and who are motivated to quit smoking. Subjects will be n=32 subjects between 18 and 65 years of age who meet DSM-IV criteria for bipolar disorder (either Type I or II), and nicotine dependence, and smoke at least 15 cigarettes per day, with an FTND score at baseline >5, expired breath CO >10, and plasma cotinine >150 ng/ml, and are motivated to quit smoking within thirty days of the initial intake. Subjects must be on a stable dose of a mood stabilizer (e.g. lithium, valproate, carbamezepine, topiramate, gabapentin or atypical antipsychotic), and be in complete remission from active manic or hypomanic and psychotic symptoms as judged by a psychiatric evaluation. Subjects will be recruited through outpatient departments at Connecticut Mental Health Center (CMHC) and its satellite clinics. Study medications will be given for 9 weeks duration, beginning at 1 week prior to the "quit date". Bupropion [as the intermediate-release (IR) formulation] will begin at 75 mg po qd x 3days, then increase to 150 mg [as bupropion SR formulation] qd x 4 days, and then increased to a final dose of up to 150 mg po bid (300 mg/day) by Day 15 (the target quit date; TQD) as tolerated, and this dose will be continued for an additional eight (8) weeks at up to 150 mg po bid. We will allow flexible dosing above 150 mg/day to allow for adjustments needed if a bipolar subject does not tolerate the full dose of Zyban at 300 mg/day. Zyban will then be discontinued at the end of Week 10. Primary outcome measures are endpoint (7-day) smoking abstinence and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. SCID for DSM-IV diagnoses of bipolar I or bipolar II disorder, and nicotine dependence.
2. Young Mania Rating Scale Total Score <12 at study entry.
3. BPRS Total Score < 20 at study entry
4. HAM-D 17-Item Score >12 and <25 at study entry. NB: We have set an upper limit for allowable HAM-D 17-item scores since higher scores would typically trigger the initiation of an antidepressant trial, and this study involves a placebo-controlled augmentation of existing medication therapies with bupropion.
5. Fagerstrom Test for Nicotine Dependence (FTND) score of 4 or more.
6. Smoking at least 15 cigarettes per day, and have expired breath CO level >10 ppm and plasma cotinine level >150 ng/ml at baseline.
7. Be on a stable dose of a mood stabilizer for at least 1 month (e.g. lithium, valproate, carbamazepine, atypical antipsychotic) as judged by the study psychiatrists (T. George, M.D. and H. Blumberg, M.D.), and judged by well-trained trained psychiatric clinicians (e.g. J. Vessicchio, M.S.W. or K. Sacco, Psy.D.) to be in remission from active manic, hypomanic, major depression and psychotic symptoms based on a clinical interview and SCID-IV.
8. Be able to provide informed consent to participate in this study as judged by clinical evaluation, and scoring at least 80% on a post-consent "test".

Exclusion Criteria:

1. Meet criteria for current abuse or dependence for any other alcohol or illicit substance within the past 3 months of study enrollment.
2. Current evidence by SCID-IV and clinical evaluation of suicidality, homocidality or psychosis.
3. Meet DSM-IV criteria for current major depression at the time of baseline evaluation.
4. A history of hypersensitivity or other known adverse reactions (e.g. hyperstimulation, severe agitation) to bupropion.
5. Any serious documented medical disorders which might be contraindicated with bupropion (i.e. anorexia or bulimia nervosa, history of seizure disorder, history of major head injury with loss of consciousness for a period greater than five minutes), or if the results of psychiatric/medical screening suggest reason concern of a trial of bupropion (e.g., a history of severe cardiac, renal or hepatic disease, diabetes mellitus or thyroid abnormalities which in the opinion of the study internist Dr. Lynn Sullivan would preclude participation in this study).
6. Evidence of clinically significant EKG abnormalities as judged by the study internist, Lynn E. Sullivan, M.D. (Department of Internal Medicine, YUSM), or her designate.
7. Prescription of monoamine oxidase inhibitors or the Wellbutrin® formulation of bupropion.
8. The presence of manic, mixed manic or hypomanic symptoms in the past one (1) month prior to study enrollment.
9. A lifetime history of antidepressant-induced mania or hypomania.
10. A history of suicidal ideation while taking antidepressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | End of Trial

SECONDARY OUTCOMES:
Smoking abstinence [7-day point prevalence at end of trial (EOT)] | End of Trial (7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Tony P. George, M.D., FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States